CLINICAL TRIAL: NCT04989452
Title: A Pilot Study for the Collection of Vocalized, Individual Digital Cough Sound Recordings to Understand COVID-19-like Symptom Progression
Brief Title: Cough Sound Recordings to Understand COVID-19-like Symptom Progression to Understand COVID-19-like Symptom Progression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ResApp Health Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 21002
Record Dates: First submitted 2021-07-30; First posted 2021-08-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Recordings of cough sounds from adults — Smartphone recordings of the cough sounds of participants who enrol in the study and obtain a COVID-19 rt-qPCR result.

SUMMARY:
Decentralized clinical study designed to collect further cough sounds, self-reported symptoms, and medical treatment questionnaires from participants enrolled on the COVID-Cough Study ("Study 1").

The aim of this further data collection study ("Study 2") is to:

1. develop an understanding of changes in cough sounds associated with COVID-19 and how they alter during the disease;
2. develop an understanding of other causes of COVID-19-like symptoms and their associated cough sound patterns; and
3. gain a broader understanding of the clinical outcomes of individuals who present for COVID-19 testing.

DETAILED DESCRIPTION:
This study is designed to be administered in a decentralized manner to collect self-reported COVID-19 symptoms, cough sample recordings and descriptions of recent medical treatment to investigate the following:

1. Whether patterns unique to COVID-19 disease can be detected in cough sounds collected over time;
2. The incidence of COVID-19 and other lung diseases within individuals who test negative for COVID-19;
3. Whether existing machine learning algorithms can detect the presence of disease in the lower respiratory tract in participants; and
4. Whether distinct cough sound patterns in COVID-19 disease are associated with the requirement of medical treatment for COVID-19 disease. Through the administration of Study 1, a list of potential participants will be created for whom the result of a recent rt-qPCR COVID-19 test is known. Participants have been consented to allow for outreach regarding further studies. Cough samples and answers to medical questions have been collected from these individuals at the time of testing, and the aim of Study 2 is to gather further cough samples and questionnaire answers over a period of 25 days.

ELIGIBILITY:
Inclusion Criteria:

* be aged 21 years and older;
* be a resident of the USA;
* have a personal (i.e., not shared) iPhone 6s or newer running iOS 14 or later;
* be able to read and understand English;
* be able to provide informed consent;
* be willing to follow study procedures;
* be able to provide at least 5 coughs (voluntary and/or spontaneous);
* have enrolled in the COVID-Cough Study and successfully returned an at-home rt-qPCR test to the study partner laboratory

Exclusion Criteria:

Participant has one or more medical contraindication to voluntary cough, including the following:

* Severe respiratory distress;
* History of pneumothorax;
* Eye, chest, or abdominal surgery within 3 months of enrolling for the study; or
* Hemoptysis (coughing up of blood) within 1 month of enrolling for the study;

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A list of COVID-19 positive and negative participants, and their consent to inform them of this study (and possible future studies) will be created through the administration of Study 1. Using this list of potential study participants we seek to enroll as many participants identified through Study 1 as possible (up to 1,500 individuals). Participants will be aged 21 years and older and will not be excluded based on gender, demographic group, or geographic location within the US.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Collection of cough sound audio recordings made using a smartphone, self-reported respiratory symptoms, COVID-19 rt-qPCR result and medical treatment information on 3 occasions (day 1, day 10, day 25). | 6 months
Sensitivity and specificity of using cough sound analysis on longitudinal cough sounds to detect COVID-19 as compared to rt-qPCR test. | 10 months
Sensitivity and specificity of longitudinal cough sounds to detect whether study participants have required recent medical care for COVID-19 related illness. | 10 months

SECONDARY OUTCOMES:
Confusion matrix outputs of cough sound algorithm prediction of COVID-19 severity compared against COVID-19 severity measured by a combination of medical history survey and rt-qPCR test. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Shrawan Patel, MBBS,BSc, Principal Investigator — Strategy Health
Locations (1):
- Strategy Health LLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.